CLINICAL TRIAL: NCT04063527
Title: Randomized Phase III Trial of the Need for Adjuvant Chemotherapy in Stage I Epithelial Ovarian Cancer After Comprehensive Staging Surgery
Brief Title: Phase III Trial of Stage I Ovarian Cancer After Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Japanese Gynecologic Oncology Group (Other)
Collaborators: Korean Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JGOG3020
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Epithelial Ovarian Cancer
Keywords: epithelial ovarian cancer; FIGO stage I; staging surgery; adjuvant chemotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Chemotherapy, Adjuvant; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy (Active Comparator): combination of paclitaxel and carboplatin
  Interventions: Drug: adjuvant chemotherapy
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: adjuvant chemotherapy — combination of paclitaxel and carboplatin
  Other Names: paclitaxel and carboplatin
  Arms: Standard therapy

SUMMARY:
To compare the Overall survival of adjuvant chemotherapy versus observation in stage I epithelial ovarian cancer after comprehensive staging surgery

DETAILED DESCRIPTION:
Based on the following adjustment factors, patients will be randomly assigned in a 1:1 ratio to adjuvant chemotherapy or observation groups.

1. Histologic type: clear cell adenocarcinoma/mucinous adenocarcinoma vs. serous adenocarcinoma/other histologic types
2. Facility where a subject is enrolled
3. International Federation of Gynecology and Obstetrics(FIGO) clinical staging: Stage Ia/ Ib vs. Stage Ic(b)

Group A: adjuvant chemotherapy group (standard treatment group):

While one of the following treatments will be performed, the number of cycles is entrusted to the treatment policy of each facility.

Paclitaxel plus Carboplatin (TC) therapy; Paclitaxel (PTX) 175 mg/m2 + Carboplatin(CBDCA) area under curve(AUC) 6 q3weeks day1, 3 to 6 cycles Docetaxel plus Carboplatin (DC) therapy; Docetaxel(DTX) 70 mg/m2 + CBDCA AUC 6 q3weeks day1, 3 to 6 cycles

After the start of TC therapy, switching from PTX to DTX due to an adverse event is permitted.

Group B: observation group (study treatment group): Observation only, no adjuvant chemotherapy administered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of histopathologically epithelial ovarian cancer
2. FIGO Stages Ia(Grade2/3, clear cell carcinoma), Ib(Grade2/3, clear cell carcinoma) and Ic(b)(all degree of differentiation and all histologic type)
3. Patients with a diagnosis of advanced stage by comprehensive staging or restaging laparotomy.
4. Patients who received comprehensive staging surgery (basic surgical techniques (total hysterectomy, bilateral salpingo-oophorectomy, and omentectomy) as well as peritoneal cytology, multiple biopsies of the peritoneum ([Peritoneal biopsy] see details below), retroperitoneal lymph node dissection (see details below [Retroperitoneal lymph node dissection]).

   However, for the following cases, it is eligible as a condition to record on the official document.
   * Peritoneal biopsy: peritoneal metastasis is not recognized by macroscopic and palpation in the stipulated site, and the case that biopsy has not been performed.
   * Retroperitoneal lymph node dissection: the case that lymph nodes of the stipulated range has been dissected however the prescribed number has not been reached.
5. Age: 20 or older
6. Performance status (PS):0-1
7. Case with initial therapy for postoperative primary lesion
8. Patient possible to receive the first study treatment within 8 weeks after the comprehensive staging surgery
9. Reasonable organ function
10. Patient must have signed informed consent.

Exclusion Criteria:

1. FIGO Stages Ic(a), Ic(1) and Ic(2)
2. Patients containing sarcoma elements
3. Patients with any signs of interstitial pneumonia or pulmonary fibrosis by chest radiography and CT
4. Patients with serious complications
5. Patients with active infection
6. Patients with intestinal paralysis or intestinal obstruction
7. Patients who have a synchronous malignancy or who have been progression-free less than 5 years for a metachronous malignancy
8. Patients with previous chemotherapy or radiation therapy
9. Patients with serious drug hypersensitivity
10. Patients with peripheral motor/sensory neuropathy [grade2,3,4 Common Terminology Criteria for Adverse Events (CTCAE) 4.0]
11. Patients who have had a hypersensitivity reaction to polyoxyethylated or hydrogenated castor oil
12. Patients with positive HBsAg. Patients with more than 2.1 log/copies ml based on fixed Hepatitis B virus (HBV)-DNA who are positive with either antigen-positive Hepatitis B (HBs), anti-hepatitis B core antigen or anti-hepatitis B surface antigen.
13. Patients who are inappropriate to enter this study with any safety reasons, judged by the treating physician

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2012-07-20 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 60 months
  1. In surviving patients, cut off will be on the last date the patient is confirmed to be alive.
  2. If a patient is lost to follow-up, cut off will be on the last date the patient is confirmed to be alive before being lost to follow-up.

SECONDARY OUTCOMES:
Relapse-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  1. If relapse is diagnosed through imaging, it is considered an event on the "test date" on which a "definite diagnosis" is obtained and not the test date that showed a "suspected relapse on an image." If a relapse is clinically diagnosed, not just through imaging, it is considered an event on the date on which relapse is diagnosed.
  2. Progression observed by CA-125 only shall not be handled as an event in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Tanabe, M.D., Study Chair — National Cancer Center Hospital East
Locations (103):
- Japan (98):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Tosei General Hospital, Seto-shi, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Hirosaki University School of Medicine & Hospital, Hirosaki-shi, Aomori
  - The Jikei University School of Medicine Kashiwa Hospital, Kashiwa-shi, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Ehime University Hospital, Onsen-gun, Ehime
  - Kyusyu Medical Center, Fukuoka, Fukuoka
  - Kyusyu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - JA Hiroshima General Hospital, Hatsukaichi-shi, Hiroshima
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Miyoshi Central Hospital, Miyoshi-shi, Hiroshima
  - Hospital Hakodate Hokkaido, Hakodate-shi, Hokkaido
  - JA Sapporo-Kosei general Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospita, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Kansai Rosai Hospital, Amagasaki-shi, Hyōgo
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagoshima University Medical And Dental Hospital, Kagoshima, Kagoshima-ken
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - St.Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama Minami Kyosai Hospital, Yokohama, Kanagawa
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kobe City Medical Center General Hospital, Kobe, Kobe
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto, Kyoto
  - Ise Red Cross Hospital, Ise-shi, Mie-ken
  - JA Matsuzaka Central Hospital, Matsuzaka, Mie-ken
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Aichi Cancer Center, Nagoya, Nagoya
  - Nara Prefecture General Medical Center, Nara, Nara
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Oita University Hospital, Yufu, Oita Prefecture
  - Hospital University of the Ryukyus, Nakagami-gun, Okinawa
  - Tomishiro Central Hospital, Tomishiro-shi, Okinawa
  - Okinawa Prefectural Chubu Hospital, Uruma, Okinawa
  - Kaizuka City Hospital, Kaizuka, Osaka
  - Osaka International Cancer Center, Osaka, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Kindai University Hospital, Ōsaka-sayama-shi, Osaka
  - Sakai City Medical Center, Sakai, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Koshigaya Municipal Hospital, Koshigaya-shi, Saitama
  - Dokkyo Medical University Saitama Medical Center, Koshigaya-shi, Saitama
  - Saitama Cancer Center, Shinden, Saitama
  - National Defense Medical College Hospital, Tokorozawa-shi, Saitama
  - Saitama National Hospital, Wako, Saitama
  - Sapporo Medical University Hospital, Sapporo, Sapporo
  - Shikoku Cancer Center, Matsuyama, Shikoku
  - Shimane University Hospital, Izumo, Shimane
  - Shizuoka Cancer Center, Nagaizumi-chō, Shizuoka
  - Japanese Red Cross Shizuoka Hospital, Shizuoka, Shizuoka
  - Dokkyo Medical University Hospital, Mibu, Tochgi
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokyo Women's Medical University Medical Center East, Arakawa City, Tokyo
  - Tokyo Medical And Dental University University Hospital of Medicine, Bunkyō-Ku, Tokyo
  - Nippon Medical School Hospital, Bunkyō-Ku, Tokyo
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyō-Ku, Tokyo
  - Sasaki Faundation Kyoundo Hospital, Chiyoda City, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Fuchu-shi, Tokyo
  - The Jikei University Katsushika Medical Center, Katsushika-ku, Tokyo
  - The Jikei University Daisan Hospital, Komae-shi, Tokyo
  - The Cancer Institute Hospital, Koto-Ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - Kosei General Hospital, Suginami, Tokyo
  - Tachikawa Hospital, Tachikawa-shi, Tokyo
  - Tottori Prefectural Central Hospital, Tottori-shi, Tottori
  - Tottori University Hospital, Yonago-shi, Tottori
  - Yamagata University Hospital, Yamagata, Yamagata
  - Tokuyama Central Hospital, Shunan-shi, Yamaguchi
  - Yamaguchi Red Cross Hospital, Yamaguchi, Yamaguchi
  - Nagano Municipal Hospital, Nagano
  - Saiseikai Nagasaki Hospital, Nagasaki
  - Saga University Hospital, Saga
  - Jichi Medical University Saitama Medical Center, Saitama
- South Korea (5):
  - National Cancer Center, Ilsandong, Goyang
  - Gachon University Gil Medical Center, Namdong, Incheon
  - Seoul ST' Mary's Hospital, Seocho, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul